CLINICAL TRIAL: NCT00410293
Title: NT-proBNP Testing in Patients Presenting to the Emergency Department With Acute Dyspnea: Evaluation of Effects on Treatment, Hospitalisation Rate and Costs
Brief Title: NT-proBNP in Acute Dyspnea: Effects on Treatment, Hospitalisation and Costs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: MEC-2004-201
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2006-12-12 (Estimated); Status verified 2006-12

CONDITIONS: Heart Failure; Dyspnea
Keywords: Heart failure; Diagnostic; Natriuretic peptide; NT-pro B-type natriuretic peptide; Length of stay; Costs
MeSH Terms: conditions — Heart Failure; Dyspnea; Disease

INTERVENTIONS:
Procedure: NT-proBNP testing

SUMMARY:
Diagnostic uncertainty in patients with complaints of shortness of breath presenting to the Emergency Department of a hospital may delay treatment and proper care. In patients with shortness of breath due to heart failure increased plasma levels of NT-pro-B-type natriuretic peptide (NT-proBNP) can be demonstrated. The use of NT-proBNP as a biomarker for heart failure in patients presenting to the emergency department with dyspnea might improve care and reduce length of hospital stay.

To investigate the effect of NT-proBNP testing on patient care and time to discharge the NT-proBNP test will be randomized. In patients in the study group, the NT-proBNP plasma level is determined at admission and the physician in charge will immediately receive the result of the test. In patients in the control group blood will be sampled but the physician will recieve no information on the NT-proBNP plasma level.

In our study we will investigate the effect of introduction of NT-proBNP as biomarker for heart failure on treatment, time to discharge and costs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Acute dyspnea as their most prominent complaint

Exclusion Criteria:

* Acute dyspnea due to a trauma
* Acute dyspnea due to cardiogenic shock
* Renal failure requiring dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-12; Study Completion 2006-08

PRIMARY OUTCOMES:
Time to discharge
Cost of treatment

SECONDARY OUTCOMES:
Duration of stay at the ED
Proportion of patients admitted to the hospital
Proportion of patients admitted to an intensive or coronary care unit
Specialist consultations
Medical treatment
Diagnostic investigations

CONTACTS AND LOCATIONS:
Overall Officials: Anton H. van den Meiracker, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands